CLINICAL TRIAL: NCT00085995
Title: Progression of Spinal Fusion in Ankylosing Spondylitis
Status: Completed | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040205; 04-AR-0205
Record Dates: First submitted 2004-06-18; First posted 2004-06-21 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-12-18

CONDITIONS: Ankylosing Spondylitis
Keywords: Syndesmophyte; Natural History; Ankylosing Spondylitis; AS; Spondyloarthropathy; Spondyloarthritis
MeSH Terms: conditions — Spondylitis, Ankylosing; Spondylarthropathies; Spondylarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will evaluate: 1) whether computed tomography (CT) scanning is better than regular x-rays for measuring changes in the stiffness, or fusion, of the spine in patients with ankylosing spondylitis; and 2) if CT can be used to determine how fast extra bone forms in the spine of these patients. Better ways to measure spinal fusion are needed to be able to evaluate the effectiveness of medicines in slowing or stopping its progression. CT uses x-rays to provide detailed pictures of the inside of the body and are valuable for detecting spinal abnormalities because of the precision with which it can show these structures. For the procedure, the patient lies on a table that moves into a large, donut-shaped scanner that can move around the body to take pictures at different angles, which are viewed on a computer monitor.

Patients 18 years of age and older with ankylosing spondylitis who are not currently taking or planning to receive treatment with anti-TNF alpha medications (etanercept, infliximab, adalimumab) for 1 year may be eligible for this study. Participants have eight clinic visits, scheduled at study entry and at 4, 8, 12, 16, 20, 24, and 48 months, at the NIH Clinical Center for the following procedures:

* Clinical assessment (all visits) - includes medical history and physical examination, measurement of spine flexibility with a tape measure and protractor, symptoms questionnaire
* Blood tests for measures of inflammation, including red blood cell sedimentation rate and C-reactive protein level (all visits)
* Urine pregnancy test in women of child-bearing age (visits 1, 4, 7, 8)
* X-rays of the pelvis, low back, and neck (visits 1, 4, 7)
* X-ray of the low back (visit 8)
* CT scan of the low back (visits 1, 4, 7)
* Magnetic resonance imaging (MRI) of the low back (visits 1, 4) - MRI combines a powerful magnet with an advanced computer system and radio waves to produce accurate, detailed pictures of organs and tissues. The patient lies on a table in a narrow cylinder containing a magnetic field, wearing earplugs to muffle loud noises that occur with electrical switching of the magnetic fields. He or she can speak with a staff member via an intercom system at all times during the procedure. During the scan, a contrast dye (gadolinium) is injected into the bloodstream through a catheter (plastic tube inserted in a vein) to brighten the images.

In addition, participants will complete a symptoms questionnaire by mail every 4 months for 2 years between visits 7 and 8.

...

DETAILED DESCRIPTION:
Spinal fusion is the clinical, radiological, and pathological hallmark of ankylosing spondylitis (AS). However, spinal fusion occurs slowly in AS. Serial radiographs rarely show changes over 2 years, and often 5 or more years are needed to demonstrate progression of spinal fusion. Methods that are more sensitive to changes in the extent of spinal fusion than plain radiographs are needed to test if any treatments can slow or halt spinal fusion in AS. The need for an improved measure of spinal fusion is heightened now that several new medications are available that have the potential to markedly decrease spinal inflammation in AS.

The goal of this pilot study is to test whether measurement of bone mineral density, bone volume, or bone mass at the annulus fibrosis of lumbar disc spaces by computed tomography (CT) can provide a reliable, valid, and sensitive measure of spinal fusion in patients with AS. Fifty-five participants will have lumbar spine CT scans at baseline, 12 months, and 24 months, lumbar spine magnetic resonance imaging at baseline and 12 months, and spinal radiographs at baseline, 12 months, 24 months, and 48 months. In addition, clinical assessments will be done every 4 months during the first 24 months. An option to perform only the baseline studies is also possible. No treatment is provided in the protocol. Reliability of image processing will be tested on repeated measurements of baseline scans. Reliability will also be assessed with repeat CT scans on up to 10 participants. Construct validity will be tested by correlation of CT measures with scores of plain radiographs, lumbar magnetic resonance imaging, and spinal range of motion. The sensitivity to change of the CT measures over 12 months and 24 months will be compared to those of two scoring systems based on plain radiographs.

ELIGIBILITY:
* A. LONGITUDINAL STUDY PROTOCOL:

Fifty-five patients will be studied.

INCLUSION CRITERIA:

1. Age 18 years or older
2. Diagnosis of AS by the modified New York criteria
3. Lumbar spine BASRI score of 0, 1, 2, or 3

We will aim to recruit at least 6 patients in each of the following BASRI lumbar spine categories:

* 0 or 1 (normal or suspicious changes)
* 2 (erosions, sclerosis or squaring with or without syndesmophytes or 2 or fewer vertebrae)
* 3 (syndesmophytes on 3 or more vertebrae with fusion of at most 2 vertebrae)

EXCLUSION CRITERIA:

1. Inability to provide informed consent.
2. BASRI lumbar spine score of 4 (complete fusion; 12)
3. Contraindication to MRI scanning based on the NMR Center MRI Safety Screening Questionnaire or size or weight limitations of the scanner.
4. History of allergic reactions to gadolinium-DPTA contrast used for MRI
5. Anticipated unavailability for follow-up over 2 years
6. Pregnancy
7. Onset of AS at age 16 or younger
8. Spondyloarthropathy other than AS
9. Severe scoliosis or other spinal malalignment that would complicate scan interpretation

B. CROSS-SECTIONAL (RELIABILITY) STUDY PROTOCOL

Up to 35 patients will be studied.

INCLUSION CRITERIA:

1. Age 18 years or older
2. Diagnosis of AS by the modified New York criteria (5)

EXCLUSION CRITERIA:

1. Inability to provide informed consent
2. BASRI lumbar spine score of 4 (complete fusion)<TAB>
3. Pregnancy
4. Onset of AS at age 16 or younger
5. Spondyloarthropathy other than AS
6. Severe scoliosis or other spinal malalignment that would complicate scan interpretation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: clinical sample
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2004-12-03 (Actual)

PRIMARY OUTCOMES:
Syndesmophyte growth | 1 and 2 years
  syndesmophyte growth by CT

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Colbert, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
not yet known

REFERENCES:
- [Background] Keaveny TM. Biomechanical computed tomography-noninvasive bone strength analysis using clinical computed tomography scans. Ann N Y Acad Sci. 2010 Mar;1192:57-65. doi: 10.1111/j.1749-6632.2009.05348.x. PMID 20392218
- [Background] Simkin PA, Downey DJ, Kilcoyne RF. Apophyseal arthritis limits lumbar motion in patients with ankylosing spondylitis. Arthritis Rheum. 1988 Jun;31(6):798-802. doi: 10.1002/art.1780310617. PMID 3382452
- [Background] Cann CE, Genant HK, Kolb FO, Ettinger B. Quantitative computed tomography for prediction of vertebral fracture risk. Bone. 1985;6(1):1-7. doi: 10.1016/8756-3282(85)90399-0. PMID 3994856
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2004-AR-0205.html